CLINICAL TRIAL: NCT01679652
Title: The Effects of Nebivolol on the NO-system in Patients With Essential
Brief Title: The Effects of Nebivolol on the NO-system in Patients With Essential Hypertension
Acronym: NEBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, MD, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHC-1-2012
Record Dates: First submitted 2012-09-01; First posted 2012-09-06 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; Nitric oxide; Nebivolol; Fractional excretion of sodium
MeSH Terms: conditions — Essential Hypertension | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebivolol (Experimental): Tablet Nebivolol 5 mg (oral use) for 5 days
  Interventions: Drug: Nebivolol
- Placebo (Placebo Comparator): Inactive placebo given as tablet for 5 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Nebivolol — Tablet i blinded in capsula
  Other Names: Tradename in Denmark: Hypoloc
  Arms: Nebivolol
Drug: placebo
  Arms: Placebo

SUMMARY:
Investigators want investigate the following hypothesis:

1. Nebivolol increases nitric oxide activity in the systemic circulation and the kidney
2. The increased activity of nitric oxide during nebivolol treatment can be demonstrated by inhibition of NO synthesis with L-NMMA. We expect increased responses in blood pressure and sodium excretion is expected during nebivolol treatment compared to placebo.

DETAILED DESCRIPTION:
Beta-blockers are no longer recommended as first line treatment in essential hypertension. Evidence mainly based on clinical trails with the non-vasodilating beta-blockers atenolol and propanolol points towards that beta-blockers have an increased risk of stroke compared to ACE-inhibitors, calcium channel blockers and thiazides. However, this Nebivolol is a third generation beta-blocker with vasodilating properties. Nebivolol decreases peripheral blood pressure to the same extend as other beta-blockers but in contrast to atenolol nebivolol also reduces central blood pressure. Furthermore nebivolol increases nitric oxide (NO) availability in forearm vessels, maybe through activation of beta-3 receptors. The nitric oxide system plays a central role in both renal sodium and water handling and regulation of vascular tone and blood pressure. It has not been investigated if nebivolol changes NO availability in the kidney.

Investigators want investigate the following hypothesis:

1. Nebivolol increases nitric oxide activity in the systemic circulation and the kidney
2. The increased activity of nitric oxide during nebivolol treatment can be demonstrated by inhibition of NO synthesis with L-NMMA. Investigators expect increased responses in blood pressure and sodium excretion is expected during nebivolol treatment compared to placebo.

Purpose The purpose of this study is to investigate the effects of nebivolol on renal handling of sodium and water (Glomerular filtration rate, urine production, free water clearance, excretion of proteins from epithelial sodium channels (u-ENaCαβγ) and aquaporin channels (u-AQP2) and sodium and potassium excretion), plasma concentrations of vasoactive hormones (renin, angiotensin II, aldosterone, vasopressin, atrial natriuretic peptide, brain natriuretic peptide and endothelin), central blood pressure, pulse wave velocity (PWV) and augmentation index, under basal conditions and during inhibition of nitric oxide synthesis in patients with essential hypertension.

Design 25 patients with essential hypertension are recruited in this randomised, cross over, placebo-controlled, double blinded study with two treatment periods (nebivolol/placebo). Each subject will attend to two examination days. Four days prior to each examination days and on the morning of each examination day subjects are given either nebivolol 5 mg pr. day or placebo. During treatment periods subject are given a standardized diet. On the examination days subject are given L-NMMA, a nitric oxide synthase inhibitor, and renal function, central hemodynamic and vasoactive hormones are evaluated during basal conditions and during inhibition of nitric oxide synthesis.

Perspectives This study is expected to contribute to increasing the knowledge about the mechanisms involved in the development and progression of cardiovascular disease. Beta-blockers are not recommended as first line treatment in essential hypertension but the results from this study may influence clinical treatment of essential hypertension in the future.

ELIGIBILITY:
Inclusion Criteria:

* Increased blood pressure (above 135 mmHg systolic or 85 mmHg diastolic in day time in 24 hour blood pressure measurement taking 5 or 10 mg amlodipine
* Men and women
* age 40 - 70 years
* informed consent

Exclusion Criteria:

* diabetes mellitus
* glomerular filtration rate < 30 ml/min
* albuminuria > 1,5 g/l
* renogram which suggests secondary hypertension
* clinical signs of pheochromocytoma or increased p-metanephrines
* clinical important sign og heart, lung, liver, thyroid or neoplastic diseases
* clinical important deviations in routine blood samples or ECG
* drug or alcohol abuse
* pregnancy or nursery
* intolerance to nebivolol
* blood donation with a month of the first examination day
* inacceptable increase in blood pressure durin L-NMMA infusion (200/120)
* inacceptable side effects to amlodipine
* blood pressure increase above 170/105 on highest dose amlodipine (10 mg)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Fractional excretion of sodium | 5 days

SECONDARY OUTCOMES:
Blood pressure | 5 days
  Both ambulatory blood pressure and office and central blood pressure before and during L-NMMA infusion
Pulse wave velocity | 5 days
  before and during L-NMMA infusion
Plasma renin concentration | 5 days
  before and during L-NMMA infusion
Plasma aldosterone concentration | 5 days
  Before and during L-NMMA infusion
Plasma angiotensin II concentration | 5 days
  Before and during L-NMMA infusion
Plasma Endothelin concentration | 5 days
  Before and during L-NMMA infusion
Plasma brain natriuretic peptide concentration | 5 days
  Before and during L-NMMA infusion
Plasma vasopressin concentration | 5 days
  Before and during L-NMMA infusion
Glomerular filtration rate | 5 days
  Before and during L-NMMA infusion
Urinary excretions of epithelial sodium channels | 5 days
  Before and during L-NMMA infusion
Urinary excretions of aquaprorin-2 | 5 days
  Before and during L-NMMA infusion
24-hour ambulatory blood pressure | 5 days
Free water clearance | 5 days
  Before and during L-NMMA infusion
Urine flow | 5 days
  Before and during L-NMMA infusion

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, MD, Study Chair — Department of medical Research, Holstebro Hospital; Frank H Mose, MD, Principal Investigator — Department of Medical Research, Holstebro Hospital
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Denmark